CLINICAL TRIAL: NCT02802566
Title: BMI-Based Prenatal Vitamins to Ameliorate Oxidative Stress in Obese Pregnancy
Brief Title: BMI-based Vitamins in Obese Pregnant Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Sarbattama Sen, Assistant Professor of Pediatrics, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2014P001393
Record Dates: First submitted 2016-05-26; First posted 2016-06-16 (Estimated); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Obesity
Keywords: Maternal Obesity; Inflammation
MeSH Terms: conditions — Obesity; Pregnancy in Obesity; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigative (Experimental): This arm receives a standard prenatal (provided by the study) and a micronutrient supplement.
  Interventions: Dietary Supplement: BMI-based prenatal vitamin
- Control (Active Comparator): Standard prenatal vitamin provided by the study
  Interventions: Dietary Supplement: Standard prenatal vitamin

INTERVENTIONS:
Dietary Supplement: BMI-based prenatal vitamin — The intervention group receives additional antioxidant micronutrients that we have found to be decreased in obese pregnant women.
  Arms: Investigative
Dietary Supplement: Standard prenatal vitamin — Standard prenatal vitamin
  Arms: Control

SUMMARY:
The purpose of this study is to devise and pilot a BMI-based prenatal vitamin for obese pregnant women. Currently, all pregnant women, regardless of body mass index, take the same prenatal vitamin. The investigators have found that obese pregnant women have higher levels of inflammation and oxidative stress, and a concomitant depletion of specific antioxidant micronutrients. The investigators have also found, in an animal model, that decreasing inflammation and oxidative stress during obese pregnancy was associated with improved offspring outcomes. Here the investigators aim to understand whether a BMI-based prenatal vitamin is effective in decreasing markers of inflammation and oxidative stress by raising concentrations of antioxidant micronutrients and in pregnancies complicated by obesity.

DETAILED DESCRIPTION:
The investigators' central hypothesis is that pregnancy in obese women creates an oxidant/anti-oxidant imbalance, which adversely impacts maternal health and neonatal outcome. The investigators hypothesize that restoring oxidant/anti-oxidant balance with a body mass index (BMI) based prenatal micronutrient supplement will decrease oxidative stress. The investigators aim to devise a prenatal vitamin supplement based on maternal BMI to increase serum levels of antioxidant vitamins in obese pregnancy, to assess how the BMI-based prenatal vitamin supplementation impacts markers of oxidative stress and inflammation in obese pregnant women and to evaluate the effectiveness of this vitamin formulation in reducing oxidative stress and inflammation and improving growth trajectories in infants born to obese women.

The investigators will conduct a double-blind randomized-controlled study. Two groups of women will be randomized independently. 1) Obese women (BMI>30) planning pregnancy through the through advertising and mailings (N=50) and 2) Pregnant women who are early in pregnancy (<13 weeks) will be approached at their first prenatal visit at the BWH and BIDMC obstetric practices (N=120).

Women will be prescreened and approached by study staff if they qualify. After informed consent is obtained, patients will be randomized to either control or intervention group by computer-generated permuted block randomization. All subjects will be given a standard prenatal vitamin provided by the study and in addition, the control group will be given a placebo and the Intervention group will be given a supplement with vitamin C, E, B6 and folate.

The outcomes are maternal systemic markers inflammation and oxidative stress and micronutrients. At the time points mentioned above, the following laboratory assays will be conducted in maternal blood or urine: C reactive protein, vitamins C, E, B6, folate 8-iso-PGF2a and 8-OHdG. The secondary outcomes are cord blood markers of inflammation and oxidative stress, breastfeeding outcomes, and the following infant outcomes over the first year: neurodevelopmental outcome, growth trajectories and adiposity, systemic markers of inflammation and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Pre-pregnancy weight or early first trimester weight (BMI > or equal to 30 kg/m2)
* Women can be either planning pregnancy (who are trying to conceive or will be trying to conceive in the coming 6 months) or <14 weeks pregnant

Exclusion Criteria:

* More than two first trimester pregnancy losses
* History of delivering an infant with a major congenital anomaly
* Pre-existing diabetes
* Autoimmune disease such as lupus
* Chronic inflammatory condition such as rheumatoid arthritis
* Uncontrolled stage two or three hypertension at baseline (systolic>160 or diastolic>100 mmHg)
* On anticoagulant therapy
* History of cigarette smoking within the past 12 months
* Lactose intolerant
* Vegan
* Unwilling to stop taking their current supplements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2014-12; Primary Completion 2017-09 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Maternal systemic marker of inflammation | 35-40 weeks of pregnancy
  Serum C Reactive Protein
Maternal systemic marker of oxidative stress | 35-40 weeks of pregnancy
  Urinary 8-Oh-dG

SECONDARY OUTCOMES:
Maternal antioxidant vitamins | 35-40 weeks of pregnancy
  Plasma Vitamin C
Maternal antioxidant vitamins | 35-40 weeks of pregnancy
  Serum Vitamin B6
Maternal antioxidant vitamins | 35-40 weeks of pregnancy
  Serum Vitamin E
Maternal antioxidant vitamins | 35-40 weeks of pregnancy
  Serum and Red Blood Cell folate
Cord blood marker of inflammation | Delivery
  Serum C Reactive Protein
Cord blood markers of oxidative stress | Delivery
  8-epi-PGF2 alpha
Breastfeeding intensity | two, six and twelve months postpartum
  Complete questionnaire on infant feeding
Infant weight | birth, 6 months and one year
  Measure infant weight (kg)
Infant length | birth, six months and one year
  length (cm) measured using a length board
Infant head circumference | birth, six months and one year
  head circumference (cm) will be measured using tape measure technique
Infant adiposity | birth, six months and one year
  adiposity by peapod measurement at birth and by skin fold thickness at birth, six months and one year
Infant marker of inflammation | 1 year
  Serum C Reactive Protein

CONTACTS AND LOCATIONS:
Overall Officials: SARBATTAMA SEN, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Non-PHI, deidentified IPD will be shared with requesting investigators. A limited data set, generated based on variables identified in an analysis plan approved by PNV investigators, will be sent via secure email or shared dropbox to requesting investigators.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be shared after publication of primary outcomes manuscript for a period of ten years.
Access Criteria: Investigators requesting access will be asked to submit a proposal and analysis plan to analyze the requested data, including plans for dissemination and authorship.

REFERENCES:
- [Background] Sen S, Simmons RA. Maternal antioxidant supplementation prevents adiposity in the offspring of Western diet-fed rats. Diabetes. 2010 Dec;59(12):3058-65. doi: 10.2337/db10-0301. Epub 2010 Sep 7. PMID 20823102
- [Background] Sen S, Iyer C, Meydani SN. Obesity during pregnancy alters maternal oxidant balance and micronutrient status. J Perinatol. 2014 Feb;34(2):105-11. doi: 10.1038/jp.2013.153. Epub 2013 Dec 19. PMID 24355940
- [Background] Panagos PG, Vishwanathan R, Penfield-Cyr A, Matthan NR, Shivappa N, Wirth MD, Hebert JR, Sen S. Breastmilk from obese mothers has pro-inflammatory properties and decreased neuroprotective factors. J Perinatol. 2016 Apr;36(4):284-90. doi: 10.1038/jp.2015.199. Epub 2016 Jan 7. PMID 26741571
- [Derived] Sen S, Cherkerzian S, Herlihy M, Hacker MR, McElrath TF, Cantonwine DE, Fichorova R, Oken E, Meydani SN. Supplementation with antioxidant micronutrients in pregnant women with obesity: a randomized controlled trial. Int J Obes (Lond). 2024 Jun;48(6):796-807. doi: 10.1038/s41366-024-01472-z. Epub 2024 Feb 23. PMID 38396126